CLINICAL TRIAL: NCT04549233
Title: The Good Tastes Study: Young Children's Response to Vegetables and Caregiver Perceptions Regarding Their Children's Food Acceptance Patterns
Brief Title: The Good Tastes Study: Young Children's Food Acceptance Patterns
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Sugar Association (Unknown); Purdue University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-2437
Record Dates: First submitted 2020-08-18; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Food Neophobia; Parenting
Keywords: Infant Feeding; Toddler Feeding; Complementary Feeding; Food Acceptance; Parenting
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children begin developing food acceptance and preferences during the first years of life, especially through repeated exposure and increased familiarity. Caregivers pay attention to the amounts of food that their children consume, and they also are sensitive to when their refuses to eat what is offered. This study will examine the interactions between caregivers and their infants when bitter vegetables are introduced to infants and toddlers. The goals for this study are to:

1. understand if masking bitterness with very low levels of sugar or salt may facilitate whether infants accept new vegetables;
2. understand if masking bitterness impacts caregivers' perceptions of infants' acceptance of new vegetables; and
3. understand the stress levels experienced by infants and caregivers throughout this process.

DETAILED DESCRIPTION:
During a single visit, four versions of a kale puree will be made with 1) no added sugar or sodium; 2) 1.2% added sugar; 3) 1.8% added sugar; and 4) 0.2% added sodium to mask bitterness. First, a familiar food will be offered to provide baseline data. Then each of the four versions of the novel kale puree will be offered to the infant by their caregiver, and the order the kale versions are presented will be randomized. The salt version will always be offered last to control for the effects of a very different taste exposure (salt vs. sweet) and to try to avoid any significant carryover effects of salt taste on sweet perception. Feeding interactions will be video recorded for behavioral coding of infant responses to each bite. Additionally, infant and caregiver heart rate and skin conductance will be monitored to assess physiological responses in each participant throughout the feeding interaction.

Several measures will be observed in order to test predictors of infant food acceptance, caregiver perceptions of infants' responses, and physiological responses in infants and caregivers. These include:

* Demographic measures
* Observed caregiver height and weight
* Observed infant length and weight
* Child developmental stage using Ages and Stages screening tool
* Caregiver neophobia
* Caregiver preferences for and intake of fruits and vegetables
* Infant feeding history and food experience
* Eating behaviors using the Child Eating Behavior Questionnaire for Toddlers
* Infant behavior using the Infant Behavior Questionnaire-Revised (Garstein & Rothbart 2003 Infant Behav Dev)
* Caregiver feeding persistence

ELIGIBILITY:
Inclusion Criteria:

* Term birth (gestational age > 37 weeks);
* Experience with at least 1 complementary food (e.g., infant cereal);
* Caregivers who are > 18 y and < 51 y of age;
* Caregivers who live within 75 miles of the University of Colorado-Denver campus.

Exclusion Criteria:

* Has genetic disorders or developmental disabilities as these conditions often result in feeding difficulties;
* Has a reported illness or metabolic disorder that would affect food intake (e.g., significant history of allergies);
* Born prematurely (< 37 weeks gestation);
* Caregivers who are younger than 18 y of age or > 51 y;
* Caregivers who live more than 75 miles from the University of Colorado-Denver campus;
* Caregivers who do not read and speak English.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and caregivers who live in the Denver area will be recruited using advertising flyers, emails sent through a university listserv and parent email distribution, and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-01-07 (Actual); Study Completion 2018-01-07 (Actual)

PRIMARY OUTCOMES:
Infant rate of acceptance of kale puree | Baseline
  Acceptance is measured using an adaptation of the Feeding Infants: Behavior and Facial Expression Coding System (FIBFECS) on a 4-point scale from 0-3 where 0 = refusal and 3 = early acceptance of food. (Hetherington et al. 2016 Food Qual Prefer)
Infant responses to kale puree | Baseline
  Responses are measured using an adaptation of the Feeding Infants: Behavior and Facial Expression Coding System (FIBFECS). Positive behaviors include leaning forward, and negative behaviors include turning head away, getting fussy, and pushing the spoon away. (Hetherington et al. 2016 Food Qual Prefer)

SECONDARY OUTCOMES:
Caregivers' perceived ratings of infant liking of kale | Baseline
  After feeding each vegetable version, the caregiver will be instructed to rate how much he/she thought his/her infant liked the vegetable using a 9-point scale ranging from 1 = "dislikes extremely", 5 = "neither likes nor dislikes", to 9 = "likes extremely"(19).
Caregivers' intentions to offer kale again | Baseline
  After feeding each vegetable version, the caregiver will be instructed to rate how likely he/she is to offer his/her infant kale in the future. Caregivers will be asked to respond using a 5-point scale ranging from 1 = "note at all likely" to 5 = "very likely".
Infant mean heart rate reactivity to kale exposure | Baseline
  Infant heart rate will be collected through disposable leads placed on the infant's torso. The mean heart rate for each of the four vegetable versions will be compared to the mean heart rate when given a familiar food.
Infant amplitude of skin conductance in response to kale exposure | Baseline
  Infant skin conductance will be collected by placing a lead on the infant's foot. The amplitude of voltage across a resistor is measured to calculate the amplitude of skin conductance. (Lykken and Venables 1971 Psychophysiology)
Caregiver mean heart rate reactivity to infant exposure to kale | Baseline
  Caregiver heart rate will be collected by placing disposable leads on the caregiver's torso. The mean heart rate recorded during the offering of each of the four vegetable versions will be compared to the mean heart rate during the offering of a familiar food.
Caregiver amplitude of skin conductance in response to infant exposure to kale | Baseline
  Caregiver skin conductance will be collected by placing a lead on the caregiver's finger.
  The amplitude of voltage across a resistor is measured to calculate the amplitude of skin conductance. (Lykken and Venables 1971 Psychophysiology)
Infant respiratory sinus arrhythmia (RSA) in response to kale exposure | Baseline
  Infant heart rate will be collected through disposable leads placed on the infant's torso. Respiratory sinus arrhythmia, the heart rate response to breathing, will be calculated using a proprietary algorithm through CardioBatch Plus (Brain-Body Center, University of North Carolina, Chapel Hill). The mean RSA observed during the offering of each vegetable version will be compared to the mean RSA observed during the offering a familiar food.
Caregiver respiratory sinus arrhythmia (RSA) in response to infant exposure to kale | Baseline
  Caregiver heart rate will be collected by placing disposable leads on the caregiver's torso. Respiratory sinus arrhythmia, the heart rate response to breathing, will be calculated using a proprietary algorithm through CardioBatch Plus (Brain-Body Center, University of North Carolina, Chapel Hill). The mean RSA observed during the offering of each vegetable version will be compared to the mean RSA observed during the offering a familiar food.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Johnson, PhD, Principal Investigator — UC Denver; Kameron J Moding, PhD, Principal Investigator — Purdue University
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available upon request to the Principal Investigator

REFERENCES:
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Squires J, Bricker D, Potter L. Revision of a parent-completed development screening tool: Ages and Stages Questionnaires. J Pediatr Psychol. 1997 Jun;22(3):313-28. doi: 10.1093/jpepsy/22.3.313. PMID 9212550
- [Background] Ham J, Tronick E. Infant resilience to the stress of the still-face: infant and maternal psychophysiology are related. Ann N Y Acad Sci. 2006 Dec;1094:297-302. doi: 10.1196/annals.1376.038. PMID 17347365
- [Derived] Johnson SL, Moding KJ, Grimm KJ, Flesher AE, Bakke AJ, Hayes JE. Infant and Toddler Responses to Bitter-Tasting Novel Vegetables: Findings from the Good Tastes Study. J Nutr. 2021 Oct 1;151(10):3240-3252. doi: 10.1093/jn/nxab198. PMID 34191021